CLINICAL TRIAL: NCT05752071
Title: GaStrointestinal STIMULation As a Treatment of Postoperative IlEus Following Extensive Surgery (STIMULATE). -A Prospective Double-blinded Randomized Controlled Trial
Brief Title: Gastrointestinal Stimulation As a Treatment of Postoperative Ileus Following Extensive Surgery
Acronym: STIMULATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: The Stimulate Study
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Ileus; Bowel Paralysis
Keywords: Stimulation; Postoperative ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment group (Experimental): A pace lead is mounted on the stomach, and exteriorized trough the skin and connected to an external pacemaker. The pacemaker is set to the following settings: 10,5 Volt, 14 hz, 330 Micro sec, Cycling 5 seconds off 0,1 sec on. The pacemaker is turned on.
  Interventions: Device: Gastric electrical stimulation
- Control group (Sham Comparator): A pace lead is mounted on the stomach, and exteriorized trough the skin and connected to an external pacemaker. The pacemaker is turned off.
  Interventions: Device: Gastric electrical stimulation

INTERVENTIONS:
Device: Gastric electrical stimulation — Mounting of a temporary gastric pacemaker

SUMMARY:
The goal of this clinical trial is to investigate the effect of gastrointestinal stimulation with a pacemaker on the length of postoperative bowel paralysis in patients undergoing major abdominal surgery due to metastasizing colorectal cancer, appendiceal cancer or pseudomyxoma peritonei.

The main question it aims to answer is if the length of postoperative ileus is reduced when the gastrointestinal tract is stimulated with a pacemaker.

All participants will undergo cytoreductive surgery +/- heated intraperitoneal chemotherapy (the standard treatment for colorectal cancer, appendiceal cancer with peritoneal carcinomatosis or pseudomyxoma peritonei). After surgery, but before the abdomen is closed a pace lead will be attached to the stomach, exteriorized trough the abdominal wall and connected to an external pacemaker. The pacemaker is either turned on (experimental group) or off (control group).

After surgery, patients will be asked to fill out a diary on bowel movements once a day. Once normal bowel function is regained, the pace lead and pacemaker will be removed trough the abdominal wall with a firm pull.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective cytoreductive surgery with or without heated intraperitoneal chemotherapy due to either colorectal or appendiceal cancer or with peritoneal metastases or due to pseudomyxoma peritonei
* Written and orally informed consent
* Over 18 years of age

Exclusion Criteria:

* Previous upper gastric or esophageal resection
* History of difficulties in swallowing or gastrointestinal stenosis
* Implanted or portable electrical medical device e.g. cardiac pacemaker, defibrillator or infusion pump etc.
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time from surgery till first stool | Approx. 7 days
  Daily patient diary information regarding stool and flatus

SECONDARY OUTCOMES:
Whole gut and regional transit times | Day of surgery til passage of SmartPill (or loss of battery ) approx. +5 days
  Measured with the SmartPill
Length of hospital stay | approx 14 days
  Number of days from primary surgery to hospital discharge
Medical complications | approx 14 days
  Any cerebral, cardiac, pulmonary, infectious, urogenital and thromboembolic complications
Surgical complications including anastomotic leakage | approx 14 days
  Surgical complications include bleeding, fascia dehiscence, mechanical ileus, surgical site infection, intraabdominal infection, anastomotic leakage
Need for surgical or radiological interventions | approx 14 days
  The number of times and the surgical or radiological procedure performed
Re-hospitalization within 30 days | From day of surgery + 30 days
  The number of re-hospitalizations and the cause of re-hospitalizations within 30 days og primary surgery
Time till initiation of postoperative systemic adjuvant chemotherapy, if indicated | From day of surgery +90 days
  In patients where indicated, the number of days fra surgery till initiation og systemic adjuvant chemotherapy
90-day mortality | From day of surgery +90 days
  Mortality within 90 days of primary surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Funder, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No